CLINICAL TRIAL: NCT01505322
Title: Persistent Pain to Impair Daily Activities Following Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kim Wildgaard, MD, Rigshospitalet, Denmark
Other Study IDs: RH2011-srv01
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Pain
Keywords: daily activities
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thoracic surgery: Lung cancer patients

SUMMARY:
Can pain impairment of daily activities be shown to be procedure specific, and thus used as an alternative to pain scoring.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years old
* Elective lung cancer surgery (VATS)

Exclusion Criteria:

* Non-Danish residence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having thoracic surgery for lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pain impairment | >12 months
  We measure persistent pain impairment in patient > 12 months folowing surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kim Wildgaard, MD, Principal Investigator — Section for Surgical Pathophysiology; Henrik Kehlet, MD, Study Director — Section for Surgical Pathophysiology
Locations (1):
- Section for Surgical Pathophysiology 4074, Copenhagen, Denmark